CLINICAL TRIAL: NCT00839228
Title: Randomised Double Blind Placebo Controlled Trial of Perhexiline in Heart Failure With Preserved Ejection Fraction Syndrome (HFpEF)
Brief Title: Perhexiline Therapy in Heart Failure With Preserved Ejection Fraction Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RRK 3147; RRK 3147 (Other: Research and Development); MREC 08/H1207/84 (Other: Ethics); EudraCT 2006-001109-28 (Registry Identifier: European Clinical Trials)
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Diastolic Heart Failure
Keywords: diastolic dysfunction; cardiac energetics; perhexiline; magnetic resonance spectroscopy
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Perhexiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perhexiline (Experimental): perhexiline 100mg o bd for 3 months
  Interventions: Drug: Perhexiline
- Placebo (Placebo Comparator): Placebo one tablet bd for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Perhexiline — 100mg o bd for 3 months
  Other Names: Pexsig
  Arms: Perhexiline
Drug: Placebo — Placebo one tablet bd for 3 months
  Other Names: Starch Placebo
  Arms: Placebo

SUMMARY:
Up to half of all patients with clinical features of heart failure are found to have normal heart pumping function. Recently the investigators have shown that a drug called perhexiline markedly improved exercise capacity and symptoms in patients with heart failure associated with impaired cardiac pump function. In this proposal the investigators will assess whether perhexiline has beneficial effects in patients with heart failure and a normal heart pumping function.

DETAILED DESCRIPTION:
Up to 50% of patients with symptoms of heart failure have a preserved left ventricular ejection fraction (HFpEF syndrome). Current therapy for systolic heart failure is targeted at inducing vasodilation and counteracting neuro-endocrine activation. There is a lack of a corresponding evidence base for the treatment of HEpEF. We have previously shown that perhexiline, an agent that increases the efficiency of energy production by shifting substrate utilization from free fatty acids towards glucose, was highly effective in improving exercise capacity, symptoms and cardiac function in patients with systolic heart failure. We have also recently shown that energy deficiency plays a major role in the pathophysiology of HFpEF. In this proposal we therefore aim to investigate the effectiveness of perhexiline in 70 HFpEF patients, in a 3 month randomised, double-blind, controlled trial. An interim analysis is planned after 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* HFpEF will be defined as:

  * Clinical features consistent with heart failure
  * LVEF ≥ 50%, with no evidence of significant valvular disease
  * No hypertrophic cardiomyopathy, and no evidence of pericardial constriction
  * Peak VO2 < 80% predicted, with RER>1 and with a pattern of gas exchange on metabolic exercise testing indicating a cardiac cause for limitation)
* Patients recruited will be in sinus rhythm

Exclusion Criteria:

* BMI >35
* Objective evidence of lung disease on formal lung function testing
* Reversible myocardial ischaemia on contrast-enhanced myocardial stress Echocardiography, and no evidence of exercise-induced mitral regurgitation (>2+)
* Impaired hepatic function; known hypersensitivity to perhexiline

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in Peak oxygen consumption (Vo2max) | 3 months

SECONDARY OUTCOMES:
Symptomatic Status (Modified Minnesota Living with Heart Failure Questionnaire) | 3 Months
Resting myocardial energetics by cardiac MR spectroscopy (MRS) | 3 months
Resting and exercise diastolic function (nuclear studies) | 3 months
Indirect measures of resting LVEDP (tissue Doppler E/Ea) | 3 months
Global LV Ejection Fraction (MRI / nuclear studies) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Frenneaux, MBBS MD, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- [Derived] Singh S, Beadle R, Cameron D, Rudd A, Bruce M, Jagpal B, Schwarz K, Brindley G, Mckiddie F, Lang C, Dawson D, Frenneaux M. Randomized double-blind placebo-controlled trial of perhexiline in heart failure with preserved ejection fraction syndrome. Future Cardiol. 2014 Nov;10(6):693-8. doi: 10.2217/fca.14.62. PMID 25495811